CLINICAL TRIAL: NCT02868268
Title: N2015-01: Neuroblastoma Precision Trial
Brief Title: Neuroblastoma Precision Trial
Status: Active, not recruiting | Type: Observational
Sponsor: New Approaches to Neuroblastoma Therapy Consortium (Other)
Collaborators: Children's Hospital Los Angeles (Other); The Evan Foundation (Other); St. Baldrick's Foundation (Other); Press On Fund (Unknown); Rising Tide Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: N2015-01; N2015-01 (Other: NANT Consortium)
Record Dates: First submitted 2016-06-03; First posted 2016-08-16 (Estimated); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood obtained (any time prior to and up to the day of biopsy) Biopsy of soft tissue, bone, bone marrow Specimens tumor content for genetic +/- IHC analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Relapsed/Refractory Neuroblastoma Pts: History of high risk neuroblastoma (NBL) according to Childrens Oncology Group (COG) risk classification with relapsed/progressive, refractory or persistent neuroblastoma. Archival or biopsied tumor specimens are provided for gene panel sequencing to subjects with potentially targetable genetic and/or immunologic biomarkers. A clinical report will be provided to subjects/subject physician detailing observed mutations and identified NBL subgroups and information on clinical trials that best match them. Subjects will be followed and data collected on treatments administered for one year after receiving this clinical report.
  Interventions: Other: Gene panel sequencing of tumor specimens

INTERVENTIONS:
Other: Gene panel sequencing of tumor specimens — Archival or biopsied tumor specimens will undergo gene panel sequencing to identify subgroups with targetable genetic (ALK, MAPK pathway, Metabolic-related genes) and/or immunologic (tumor associated macrophage infiltration, PD-L1 expression) biomarkers in neuroblastoma. A clinical report will be provided to subjects/subject physician detailing observed mutations and identified NBL subgroups and information on clinical trials that best match them. Subjects will be followed and data collected on treatments administered for one year after receipt of clinical report.

SUMMARY:
This proposal sets forth the platform for a Precision Medicine clinical trial through the New Approaches to Neuroblastoma Therapy (NANT) consortium. The plan is to utilize NANT's established multi-institutional infrastructure and Translational Genomics Research Institute GEM sequencing platform for acquisition and gene panel sequencing of relapsed biological specimens in relapsed/refractory neuroblastoma (rNB) including those obtained from the bone, bone marrow or soft tissue. Our primary aim is to identify subgroups of rNB patients who have potentially targetable genetic (ALK, MAPK pathway, Metabolic-related genes) and/or immunologic (tumor-associated macrophage infiltration and/or programmed death ligand [PD-L1] expression) biomarkers in rNB. Additional potential novel biomarkers will also be evaluated and reported in this cohort of patients.

DETAILED DESCRIPTION:
Neuroblastoma (NB) is the most common extracranial solid tumor of childhood. High-risk NB is highly lethal and responsible for over 15% of childhood cancer related deaths. The majority of patients with metastatic NB respond to upfront cytotoxic chemotherapy, yet patients who die of recurrent disease do so from tumor acquired resistance to treatment. Thus, understanding the repertoire of tumor specific genomic alterations leading to tumor progression and therapy resistance is critical to devising novel targeted therapy options for patients with recurrent or refractory (r)NB. Limited data exists regarding the genetic and immunologic predictive biomarkers in rNB, which can be used to direct targeted therapies. Another barrier to clinical implementation of genetic testing of tumor samples from children with rNB is obtaining sufficient number of tumor cells from bone marrow (BM) specimens, the most easily accessible and common site of relapse. This proposal sets forth the platform for a Precision Medicine clinical trial through the New Approaches to Neuroblastoma Therapy (NANT) consortium. The plan is to utilize NANT's established multi-institutional infrastructure and Translational Genomics Research Institute (TGen) GEMTM sequencing platform for acquisition and gene panel sequencing of relapsed biological specimens in rNB including those obtained from the bone, bone marrow or soft tissue. Our primary aim is to identify subgroups of rNB patients who have potentially targetable genetic (ALK, MAPK pathway, Metabolic-related genes) and/or immunologic (tumor-associated macrophage infiltration and/or PD-L1 expression) biomarkers in rNB. Additional potential novel biomarkers will also be evaluated and reported in this cohort of patients. This aim has immediate impact on the lives of children with rNB as it provides a clinical report to patients and their physicians detailing observed mutations and rNB subgroups and information on clinical trials that best match them. Our second aim will assess a novel method for enriching tumor cells from bone marrow aspirates containing less than 30% tumor involvement so that next generation sequencing can be performed. Our bone marrow (BM) enrichment protocol has both methodological and patient significance; 1) BM enrichment will allow a much larger group of rNB patients access to future personalized medicine trials and 2) Successful confirmation that BM enrichment can produce quality DNA for genetic analysis serves as proof of principal that this method can be used for genetic testing of BM with evidence of metastasis in other adult or pediatric solid tumors. In summary, our proposal will define the genetic and immunologic landscape of rNB and contribute to our understanding and ability to therapeutically target the dynamic alterations in tumor biology of children with rNB.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 1 year and ≤ 30 years of age at study registration
* Patients must have had a diagnosis of neuroblastoma either by histological verification of neuroblastoma and/or demonstration of tumor cells in the bone marrow with increased urinary catecholamines.
* Patients must have a history of high-risk neuroblastoma according to
* COG risk classification at the time of study registration. Patients must have at least one of the following: Recurrent/progressive disease, Refractory disease, Persistent disease
* Patient must be willing to undergo a clinically indicated biopsy and meet at least one of the following requirements: Bone biopsy, Soft tissue biopsy, Bone marrow biopsy and aspirate
* Patients must not be receiving any other anti-cancer agents or radiotherapy during the interval

Exclusion Criteria:

* Patients with disease of any major organ system that would compromise their ability to withstand biopsy procedures of soft tissue, bone and/or bone marrow.
* Patients who enroll and successfully receive a NANT Precision Report may not re-enroll at a future time.
* Patient declines participation in NANT 2004-05, the NANT Biology Study.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: High risk neuroblastoma
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2016-08-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Identify genomic alterations, whether targetable alterations are present and within 4 defined NBL subgroups or outside of these 4 defined NBL subgroups. Identify presence/absence of immunologic biomarkers common to NBL. | 6 weeks
  Archival or biopsied tumor specimens undergo gene panel sequencing and/or immunohistochemistry and a list of all genetic/immunologic alterations are identified. Was an actionable genetic alteration identified and were any of these alterations within 4 NBL specific subgroups (ALK, MAPK, Metabolic, Immune reactive) or outside of the 4 NBL specific subgroups.

SECONDARY OUTCOMES:
How many subjects are biopsied or provide available tumor that is found to be adequate for gene panel sequencing and produces a clinical report | 6 weeks
  Identify number of subjects who successfully provide tumor from either a procedure or archival sources and whether this tumor is adequate for analysis (>= 30% tumor present/specimen) as determined locally and centrally. Of these specimens that are found to be adequate and sent to the gene sequencing center, how many result in a clinical report being issued.
How many patients with bone marrow aspirates performed that contain < 30% tumor cells are able to be enriched and genetic alterations identified | 1 year
  Identify number of subjects who successfully provide tumor from either a bone marrow aspiration or archival sources and < 30% tumor present. Was tumor enrichment attempted and # of patients where enrichment was attempted and successful to allow gene sequencing and identification of genetic/immunologic alterations. Was an actionable genetic alteration identified and were any of these alterations within 4 NBL specific subgroups (ALK, MAPK, Metabolic, Immune reactive) or outside of the 4 NBL specific subgroups.

CONTACTS AND LOCATIONS:
Overall Officials: Shahab Asgharzadeh, MD, Study Chair — Children's Hospital Los Angeles
Locations (11):
- United States (11):
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Children Hospital of Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Childrens Hospital Boston, Dana-Farber Cancer Institute., Boston, Massachusetts
  - C.S Mott Children's Hospital, Ann Arbor, Michigan
  - University of North Carolina, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cook Children's Healthcare System, Fort Worth, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared with the treating investigator and the study participant.